CLINICAL TRIAL: NCT05639660
Title: Aflibercept Observational Study for the Clinical Use of PCV in China, Polycentric, Observational, Retrospective-prospective Study
Brief Title: Clinical Implication of Aflibercept in PCV Treatment in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: CAPTAIN
Record Dates: First submitted 2022-10-28; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-10

CONDITIONS: Polypoidal Choroidal Vasculopathy
Keywords: Polypoidal Choroidal Vasculopathy; Aflibercept
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aflibercept group: Single arm, Aflibercept 2.0mg/0.05ml, intravitreal injection
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — The treatment guideline recommends the 3+Q2m regimen for Aflibercept, but this study is an observational study, no intervention is made in the subjects' treatment regimen. There is no prescribed visit plan. According to the decision of the doctor and the patient according to the treatment plan, the patient needs to come to the clinic within the prescribed time window (3, 6, and 12 months) to facilitate the recording of data.

SUMMARY:
The purpose of this study is to evaluate the overall treatment characteristics and efficacy of Aflibercept in the treatment of PCV in China through a multicenter, observational, prospective-retrospective study. This study is a long-term follow-up cohort, plans to unite a total of 30 hospitals in different regions of the China to enroll 1000 PCV patients.

Main evaluation indicators: To observe the changes in visual acuity (BCVA) in PCV patients treated with Aflibercept to evaluate the effectiveness of the treatment.

DETAILED DESCRIPTION:
Primary Study Objective(s) To provide overall treatment characteristics of aflibercept in PCV treatment Secondary Study Objective(s)

1. To describe the treatment regimens of aflibercept treatment on PCV in clinical practice.
2. To evaluate effectiveness of aflibercept treatment on PCV including vision gain (BCVA) and anatomic improvement (CRT, Polyps regression, Polyps inactivity, and PED)
3. To explore the relative factors of aflibercept treatment effectiveness.
4. To describe patients' tolerance to anti-VEGF and PDT treatment.
5. To collect safety information with aflibercept treatment in a wider population setting

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, gender, unilateral or bilateral onset
2. Treatment-experienced or treatment-naïve patients diagnosed with PCV after ICGA examination
3. Signed informed consent, able to long-term follow-up
4. PCV patients previously treated with aflibercept were enrolled as retrospective cases, and PCV patients previously treated with other anti-VEGF, at least 1 month since the last treatment

Exclusion Criteria:

1. Patients with anterior segment (including iris and angle) neovascularization or neovascular glaucoma
2. Received oral or intravenous antiangiogenic drugs within 180 days prior to the screening visit
3. The study eye has a history of idiopathic or autoimmune uveitis
4. Study eyes with active ocular inflammation or evidence of infectious blepharitis, corneal inflammation, scleritis, or conjunctivitis
5. The patient has a coagulation disorder or is taking oral warfarin, Plavix (clopidogrel) and other similar anticoagulation drugs.
6. The patient is receiving treatment for severe systemic infection
7. Patients with uncontrolled blood pressure (systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg when the subject is sitting)
8. Cerebrovascular accident and/or myocardial infarction within 180 days prior to the screening visit
9. Patients with renal insufficiency undergoing renal dialysis, renal failure requiring dialysis or renal transplantation
10. The investigator believes that based on the history of other diseases, metabolic dysfunction, physical examination results or clinical laboratory results, patients have a disease or condition that will increase the risk for complications from treatment
11. Pregnant or lactating women; women of childbearing potential with positive pregnancy test results at baseline or not receiving pregnancy test; postmenopausal women must have been amenorrhea for at least 12 months to not be considered fertile
12. Participated in any drug (except vitamins and minerals) or device therapy study within 30 days prior to the screening visit
13. The patient has received other anti-VEGF therapy within 30 days
14. Other patients deemed necessary to be excluded by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed as polypoid choroidal vasculopathy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of Mean BCVA from baseline at the month 3, 6, 12 | Through study completion, 1 year
  Routine International standard visual acuity chart, best corrected visual acuity
Mean treatment pattern of aflibercept in PCV treatment | Through study completion, 1 year
  To describe the mean treatment pattern of aflibercept in PCV treatment

SECONDARY OUTCOMES:
Proportion of patients with each treatment regimen | Through study completion, 1 year
  based on different count and describe the patients' proportion
Change in CRT from baseline at month 3, 6, 12 | Through study completion, 1 year
  Non-contact intraocular pressure before and after study eye injection, study eye slit lamp, ophthalmoscopy, identify the change of CRT
Proportion of patients with complete regression of polyps at month 3, 6, 12 | Through study completion, 1 year
  color fundus photography of the research eye, study eye ICGA angiography
Proportion of patients with inactivity polyps at month 3, 6, 12 | Through study completion, 1 year
  color fundus photography of the research eye, study eye ICGA angiography
Proportion of patients with dry retina at month 3, 6 and 12 | Through study completion, 1 year
  OCT, OCTA examination, color fundus photography of the research eye
Proportion of patients with PED regression at month 3, 6 and 12 | Through study completion, 1 year
  OCT, OCTA examination
Mean of treatment interval and number of injections at month 12 | Through study completion, 1 year
  Observe and describe the treatment pattern during routine follow-up visits
Inactive polyp evaluation by OCTA at month 3, 6, 12 | Through study completion, 1 year
  OCTA examination during follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Professor, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China